CLINICAL TRIAL: NCT00007722
Title: CSP #500 - An Epidemiological Investigation Into the Occurrence of Amyotrophic Lateral Sclerosis (ALS) Among Gulf War Veterans
Brief Title: Amyotrophic Lateral Sclerosis (ALS) Gulf War Study
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency); ALS Association (Other)
Responsible Party: Oddone, Eugene - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 500
Record Dates: First submitted 2000-12-29; First posted 2001-01-01 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; amyotrophic lateral sclerosis; Gulf War Veterans
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples of blood or mouthwash were collected in veterans' homes by nurses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Recently, concern has arisen regarding a possible elevated occurrence of ALS among veterans who served in the Persian Gulf during Operations Desert Shield (August 2, 1990 - January 15, 1991), Desert Storm (January 16, 1991 - February 28, 1991) and Clean-up (March 1, 1991 - July 31, 1991). This study involves an epidemiologic investigation into the occurrence of ALS among veterans of the Gulf War. This study will further define the epidemiology of this neurological disease among younger individuals while determining whether there is a higher than expected occurrence. It will also ascertain the etiologic importance of deployment to the Persian Gulf and exposure to specific environmental factors in that geographic area. VA is leading this joint federal government epidemiologic study that also involves DoD, HHS, CDC, and academic centers of excellence in neurology, with advice from the ALS Association.

DETAILED DESCRIPTION:
Primary Objectives: To develop, through nationwide ascertainment, a comprehensive descriptive epidemiology of amyotrophic lateral sclerosis (ALS) among Gulf War veterans with particular attention to whether there is a higher than expected occurrence of ALS among deployed veterans as compared to non-deployed Gulf War veterans.

Secondary Objectives: To ascertain probable/possible etiologic factors with particular focus on the role of chemical or biologic factors in the Persian Gulf area of deployment.

Primary Outcomes: Incidence of ALS among deployed and non-deployed veterans of the Gulf War.

Intervention: N/A

Study Abstract: Recently, concern has arisen regarding a possible elevated occurrence of ALS among veterans who served in the Persian Gulf during Operations Desert Shield (August 2, 1990 - January 15, 1991), Desert Storm (January 16, 1991 - February 28, 1991) and Clean-up (March 1, 1991 - July 31, 1991). In response to this concern, a nationwide epidemiological investigation was conducted to ascertain all occurrences of ALS between August, 1990 and July, 2000 among all active duty military and mobilized Reserves, including National Guard, who served during the Gulf War period (August 2, 1990-July 31, 1991). A diagnosis of ALS was confirmed by medical record review and, as necessary, neurological examination. Risk was assessed by the age-adjusted, average, annual 10-year cumulative incidence rate. VA led this joint federal government epidemiologic study that also involved DoD, HHS, CDC, and academic centers of excellence in neurology, with advice from the ALS Association.

The study population was defined as all active duty military and mobilized reserves and National Guard who served for at least one month at any time during the Gulf War period. Mobilized reservists and members of the National Guard were those who were activated and called-up, being either deployed to S.W. Asia or "back-filling" positions of military personnel who were deployed. Deployed military personnel were those who served in the S.W. Asian theater during Operations Desert Shield and Desert Storm or the period immediately after Desert Storm or received hazardous duty pay during the Gulf War. All other individuals in the study population were classified as non-deployed, although they may have been stationed outside the U.S.

This study has as its primary component a field epidemiological investigation, involving nationwide ascertainment of ALS cases among deployed and non-deployed veterans of the Gulf War to obtain a census of ALS cases among these populations. Ascertainment of cases occurred through three avenues. The first was a search of extant VA and DoD medical databases. Second, we solicited cases from the ALS Association, other related organizations, and from VA and DoD neurology clinics. And third, we identified cases through self-referrals that resulted from national media announcements. Purported cases were verified via medical record review and, as necessary, a detailed clinical examination. For all living cases, we are collecting a sample of blood and urine for determination of ALS-relevant DNA mutations and heavy metal exposure, respectively. There is also an in-home visit that includes an interview of the patient and family members with emphasis on ascertainment of unique exposures.

Results: In this large epidemiological study, researchers supported by both the Department of VA and DoD have found preliminary evidence that veterans who served in Desert Shield-Desert Storm are nearly twice as likely as their non-deployed counterparts to develop ALS. VA is exploring options for compensating veterans who served in the Gulf and who subsequently develop ALS.

Ongoing Surveillance: The study team has implemented an ongoing surveillance system to detect future cases of ALS that develop in this veteran population. This system involves maintaining the linkages created to detect current cases. New cases will be subject to the same protocols for verification, enrollment and data collection as in the original case ascertainment study.

ELIGIBILITY:
Inclusion Criteria:

Veterans who served in the Persian Gulf during Operations Desert Shield (August 2, 1990 - January 15, 1991), Desert Storm (January 16, 1991 - February 28, 1991) and Clean-up (March 1, 1991 - July 31, 1991)

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living and deceased veterans with an ALS diagnosis who served in the military between 8/2/1990 and 7/31/1991.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2000-07; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Probability of ALS among veterans both deployed and non-deployed to the Gulf Region(8/2/1990-7/31/1991) | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Z. Oddone, MD MHSc, Study Chair — VA Medical Center
Locations (1):
- VA Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Horner RD, Grambow SC, Coffman CJ, Lindquist JH, Oddone EZ, Allen KD, Kasarskis EJ. Amyotrophic lateral sclerosis among 1991 Gulf War veterans: evidence for a time-limited outbreak. Neuroepidemiology. 2008;31(1):28-32. doi: 10.1159/000136648. Epub 2008 Jun 6. PMID 18535397
- [Result] Miranda ML, Alicia Overstreet Galeano M, Tassone E, Allen KD, Horner RD. Spatial analysis of the etiology of amyotrophic lateral sclerosis among 1991 Gulf War veterans. Neurotoxicology. 2008 Nov;29(6):964-70. doi: 10.1016/j.neuro.2008.05.005. Epub 2008 Jun 23. PMID 18573277
- [Result] Kasarskis EJ, Lindquist JH, Coffman CJ, Grambow SC, Feussner JR, Allen KD, Oddone EZ, Kamins KA, Horner RD; Als Gulf War Clinical Review Team. Clinical aspects of ALS in Gulf War veterans. Amyotroph Lateral Scler. 2009 Feb;10(1):35-41. doi: 10.1080/17482960802351029. PMID 18792848